CLINICAL TRIAL: NCT01204060
Title: Effect of Allergen Challenge on Inflammation Induced by Toll-like Receptor Stimulation in a Nasal Model.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: #10-3322
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Nasal Allergen Lipopolysaccharide Inflammation Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal allergen challenge (Active Comparator)
  Interventions: Other: Nasal allergen challenge
- Nasal placebo challenge (Placebo Comparator)
  Interventions: Other: Nasal placebo challenge

INTERVENTIONS:
Other: Nasal allergen challenge — Subjects will receive a nasal spray containing an allergen to which they are allergic
  Arms: Nasal allergen challenge
Other: Nasal placebo challenge — Subjects will receive a nasal spray with allergen diluent
  Arms: Nasal placebo challenge

SUMMARY:
Asthma is one of the most common diseases affecting about 2.5 million Canadians, and can result in reduced quality of life and difficulties with work and school. Once the disease has become established with irreversible changes in the lungs it can be very difficult to treat. Severe asthma although less common than mild asthma uses more healthcare resources.

The objective of this project is to find out how the changes in the lung develop in severe asthma. Once this is known then new treatments can be developed to prevent irreversible damage to the lungs.

Volunteers will have substances sprayed up their nose and then samples collected from their nose. Levels of proteins and cells can be measured in these samples. This will give an indication of the type of inflammation that occurs.

The usual method of investigating the changes that occur in asthma is to challenge the lungs. Samples have to then be collected from the lungs. This can be in the form of sputum which must be treated to break it down to a liquid or washed out during a camera test. These methods cause problems with measuring proteins and they are broken down or diluted. Because the nose is easily accessible samples can be obtained at many time points. Because the samples can be collected directly from the nose the problems with obtaining samples from the lung are avoided.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects over the age of 18 2 Subjects able to give written informed consent 3 Subjects able to comply with study procedures and protocol 4 Subjects with a history of allergic asthma 5 Subjects with a positive skin prick test to a common aeroallergen 6 Subjects who are otherwise healthy with no other health problems

Exclusion Criteria:

1. Subjects with a viral URTI within 2 weeks prior to screening.
2. Subjects with a TNSS> 2 at screening
3. Subjects with a structural nasal abnormality or nasal polyps on examination, a history of frequent nose bleeding, nasal surgery within the previous 3 months.
4. Subjects who are a current smoker or have a history of smoking within the previous 3 months.
5. Subjects who have used a medication that could affect responses to nasal challenge (eg corticosteroids, decongestants, anti-histamines) or any other nasally applied medication within 2 weeks prior to screening.
6. Subjects who have participated in any other clinical trials within the previous 3 months.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Level of eosinophils in nasal lavage | Assessed 4 hours after challenge

SECONDARY OUTCOMES:
Change in level of IL-4, IL-5 and IL-13 in nasal secretions | Assessed 4 hours after challenge
Change in nasal symptom score | Assessed 4 hours after challenge
Change in FIZZ1 levels in nasal tissue | Assessed 4 hours after challenge

CONTACTS AND LOCATIONS:
Overall Officials: Helen Neighbour, MB BS PhD, Principal Investigator — McMaster University
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada